CLINICAL TRIAL: NCT06767267
Title: Epidemiology of Acute Otomastoiditis in Pediatric Age: a Single-center Retrospective Prospective Observational Study
Brief Title: Epidemiology of Acute Otomastoiditis in Pediatric Age
Acronym: PAM_2022
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: PAM_2022
Record Dates: First submitted 2024-12-01; First posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2024-10

CONDITIONS: Otomastoiditis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
It was decided to conduct this study because there are no standardized guidelines. regarding the management of acute otomastoiditis. The aim of the study is to describe the epidemiology of otomastoiditis in order to outline the scientific and rational basis necessary to standardize the diagnostic and therapeutic approach to this condition in order to reduce the diagnostic delay and improve the therapeutic outcome. It also aims to evaluate the effectiveness of different treatment modalities and identify possible risk factors associated with complications.

DETAILED DESCRIPTION:
Acute otomastoiditis is the main suppurative complication of acute otitis media (OMA) and is secondary to the extension of the inflammatory process from the middle ear to the mastoid process of the temporal bone through a narrow canal, termed aditus ad antrum, which in the youngest child is more likely to be obstructed (due to the absence of pneumatization of the mastoid).1,2 Rarely, mastoiditis can occur even in the absence of signs and symptoms suggestive of OMA.3 Currently, risk factors leading to the evolution of OMA into otomastoiditis are not known in the literature, so the debate on the proper management of the single episode of otitis as a preventive strategy is still very much alive, also in light of the extreme frequency of OMA in pediatric age, its frequent self-resolution and the rarity of its complications. In particular, acute otomastoiditis remains a rare complication; in fact, it is estimated that the percentage of OMA that goes on to evolve into otomastoiditis is 0.24%.

The annual incidence of acute mastoiditis has been greatly reduced since the introduction of antibiotic therapy and is estimated to be between 1.2 and 4.2 cases per 100,000 children in industrialized countries.

Over the past decades, several scientific societies have updated guidelines for the management of OMA in order to reduce the overprescription of antibiotics and the consequent increase in drug resistance.In the latest Italian guidelines, the strategy of watchful waiting, i.e., clinical observation for the first 48-72 hours after symptom onset, has been confirmed only in children older than 2 years with mild monolateral, severe monolateral, and mild bilateral OMA. According to some authors, this treatment choice did not impact the incidence of complications, particularly otomastoiditis, but conflicting opinions exist in the literature.

In recent years, numerous studies have documented an increasing trend in the incidence of acute otomastoiditis, in particular, a study conducted from 2002 to 2013 at 25 hospitals in our country documented an increase in the annual number of acute otomastoiditis in patients older than 4 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≤14 years with an established diagnosis of acute otomastoiditis

Exclusion Criteria:

* NA

Max Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study will be offered consecutively to every patient and parent and/or guardian of patients diagnosed with established acute otomastoiditis (prospective phase) accessing the Emergency Pediatrics
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2024-03-13 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Describe the epidemiology of cases of acute otomastoiditis in the pediatric population | through study completion, an average of 1 year
  Clinical outcomes of the different treatment modalities of acute otomastoiditis will be evaluated by the percentage of patients with complications after execution of the different treatment modalities performed.

CONTACTS AND LOCATIONS:
Overall Officials: Luca Pierantoni, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero - Universitaria di Bologna, U.O. Pediatria d'Urgenza, Pronto Soccorso e Osservazione Breve ed Intensiva, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No